CLINICAL TRIAL: NCT05667597
Title: Longitudinal Follow-up of SARS-CoV-2 (COVID-19) Immunity in Immunocompromised Populations in Belgium (COVICO) in Nursing Home Residents and Staff During the Winter Season 2022-2023
Brief Title: Sars-COV-2 (COVID-19) Immunity in immunoCOmpromised Populations
Acronym: COVICO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Goossens (Other Government)
Collaborators: Université Libre de Bruxelles (Other); Institute of Tropical Medicine (Other Government); Mensura EDPB (Unknown); Erasme University Hospital (Other)
Responsible Party: Sponsor-Investigator, Maria Goossens, Coordinator observational trial unit, Sciensano
Organization: Sciensano (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P2022/474; 2022-002531-56 (EudraCT Number)
Record Dates: First submitted 2022-07-04; First posted 2022-12-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: SARS CoV 2 Infection; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Immunity, Humoral

STUDY DESIGN:
Intervention Model Description: the intervention is the blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Residents and staff from nursing homes from the previous PICOV-VAC study (Experimental)
  Interventions: Diagnostic Test: Humoral immunity
- Healthy adults from the previous REDU-VAC study (Experimental)
  Interventions: Diagnostic Test: Humoral immunity
- Kidney transplant and dialysis patients from the previous NEPHRO-VAC study (Experimental)
  Interventions: Diagnostic Test: Humoral immunity
- Lung transplant patients from the previous LUNG-VAC study (Experimental)
  Interventions: Diagnostic Test: Humoral immunity

INTERVENTIONS:
Diagnostic Test: Humoral immunity — determine binding and neutralizing antibody levels against the epidemiologically predominant SARS- CoV-2 variants of concern (VOC) and the wild type SARS-CoV-2 (Wuhan strain).

SUMMARY:
The immune response of COVID-19 vaccination was monitored and studied in the context of the previously PICOV study (P2020/424), Nephro- VAC studies (P2020/284 and P2020/312) and Lung-VAC study (P2021/182). The constant emergence of new variants of concern (VOCs), which become increasingly better at escaping infection and vaccine induced immune responses, together with waning immunity over time, warrant additional vaccination rounds. This is especially true in immunocompromised populations.

In the current study, we want to continue monitoring SARS-CoV-2 specific immunity over the next two years, encompassing several future vaccination campaigns.

DETAILED DESCRIPTION:
Background: In collaboration with several Belgian universities, hospitals and institutes, Sciensano, the Belgian Scientific Institute of Public Health, set up a consortium to facilitate and streamline the organization of COVID-19 vaccination studies primarily in immunocompromised populations. The immune response of COVID-19 vaccination was monitored and studied in the context of the previously PICOV study (P2020/424), Nephro- VAC studies (P2020/284 and P2020/312) and Lung-VAC study (P2021/182). The constant emergence of new variants of concern (VOCs), which become increasingly better at escaping infection and vaccine induced immune responses, together with waning immunity over time, warrant additional vaccination rounds. This is especially true in immunocompromised populations.

In the current study, we want to continue monitoring SARS-CoV-2 specific immunity over the next two years, encompassing several future vaccination campaigns.

Method: A non-commercial multicenter academic prospective cohort study will be conducted in immunocompromised populations and healthy adults for two years. These healthy people will be recruited from the previously organized PICOV-VAC study (members of nursing home staff) (EudraCT 2021-000401-24) and REDU-VAC study (EudraCT 2021-002088-23) while the immunocompromised participants will be recruited from the previously established PICOV-VAC, REDU-VAC, Lung-VAC and Nephro-VAC cohorts from which historic clinic and immunologic data is available. Participants will be sampled three times a year independently of the vaccinations which will be administered through regular channels not linked to the study itself.

Objectives: The main goal of this study is to measure levels of immunity in healthy adults and immunocompromised participants three times a year. The primary objective is to determine binding and neutralizing antibody levels against the epidemiologically predominant SARS- CoV-2 variants of concern (VOC) and the wild type SARS-CoV-2 (Wuhan strain). This will allow us to determine to which extent extra booster doses can or cannot induce more (binding) and/or better (neutralizing) antibodies to different variants as compared to peak responses achieved after previous vaccination doses and to study waning of these responses after winter periods.

Secondary objectives include studying the vaccine induced immunity in more detail. This includes the further characterization of the quality of the antibody response and the measurement of the cellular immune response, amongst others.

ELIGIBILITY:
Inclusion Criteria:

* Being a resident or member of staff in a nursing home and having participated in the previously organized PICOV-VAC study.
* Being cognitively capable to give consent to participate in the study.
* Being a healthy adults and having participated in the previous REDU-VAC study
* Being a kidney transplant or dialysis patient and having participated in the previous NEPHRO-VAC study
* Being a lung transplant patient and having participated in the previous LUNG-VAC study

Exclusion Criteria:

* Having insufficient knowledge of the Dutch or French language..
* Having a previous diagnosis of dementia and/or having a mini-mental state examination (MMSE) score < 18/30.
* Having veins which are not accessible for simple peripheral blood puncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of SARS-CoV-2 binding and neutralizing antibodies | Three times a year, during two years
  change in the concentration of binding and neutralizing antibodies against the epidemiologically predominant SARS-CoV-2 variant of concern (VOC) and the wild type SARS-CoV-2 (Wuhan strain)

SECONDARY OUTCOMES:
Maturation of specific antibody affinity to SARS-CoV-2 | Three times a year, during two years
  change in SARS-CoV-2 specific antibody affinity maturation
Levels of mucosal antibodies to SARS-CoV-2 | Three times a year, during two years
  change of the mucosal antibodies to SARS-CoV-2
Frequencies of T and B cell to SARS-CoV-2 | Three times a year, during two years
  change of SARS-CoV-2 specific cellular immunity
Levels of non-neutralizing functions of antibodies to SARS-CoV-2 | Three times a year, during two years
  change of levels the non-neutralizing functions of antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Sciensano, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
This study is part of the BelCoVac consortium. The memorandum of understanding describes the conditions of data sharing.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Result] Goossens ME, Neven KY, Pannus P, Barbezange C, Thomas I, Gucht SV, Dierick K, Schmickler MN, Verbrugghe M, Loon NV, Arien KK, Marchant A, Goriely S, Desombere I. The prior infection with SARS-CoV-2 study (PICOV) in nursing home residents and staff - study protocol description and presentation of preliminary findings on symptoms. Arch Public Health. 2021 Nov 11;79(1):195. doi: 10.1186/s13690-021-00715-z. PMID 34763723
- [Result] Pannus P, Neven KY, De Craeye S, Heyndrickx L, Vande Kerckhove S, Georges D, Michiels J, Francotte A, Van Den Bulcke M, Zrein M, Van Gucht S, Schmickler MN, Verbrugghe M, Matagne A, Thomas I, Dierick K, Weiner JA, Ackerman ME, Goriely S, Goossens ME, Arien KK, Desombere I, Marchant A. Poor Antibody Response to BioNTech/Pfizer Coronavirus Disease 2019 Vaccination in Severe Acute Respiratory Syndrome Coronavirus 2-Naive Residents of Nursing Homes. Clin Infect Dis. 2022 Aug 24;75(1):e695-e704. doi: 10.1093/cid/ciab998. PMID 34864935
- [Result] Kemlin D, Lemy A, Pannus P, Desombere I, Gemander N, Goossens ME, Marchant A, Le Moine A. Hybrid immunity to SARS-CoV-2 in kidney transplant recipients and hemodialysis patients. Am J Transplant. 2022 Mar;22(3):994-995. doi: 10.1111/ajt.16853. Epub 2021 Oct 1. No abstract available. PMID 34554629
- [Result] Pannus P, Depickere S, Kemlin D, Houben S, Neven KY, Heyndrickx L, Michiels J, Willems E, De Craeye S, Francotte A, Chaumont F, Olislagers V, Waegemans A, Verbrugghe M, Schmickler MN, Van Gucht S, Dierick K, Marchant A, Desombere I, Arien KK, Goossens ME. Safety and immunogenicity of a reduced dose of the BNT162b2 mRNA COVID-19 vaccine (REDU-VAC): A single blind, randomized, non-inferiority trial. PLOS Glob Public Health. 2022 Dec 20;2(12):e0001308. doi: 10.1371/journal.pgph.0001308. eCollection 2022. PMID 36962838